CLINICAL TRIAL: NCT03405090
Title: Differential Mechanisms of Dyspnea Relief in Advanced COPD: Opiates vs. Bronchodilators
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dr. Denis O'Donnell (Other)
Collaborators: Ontario Lung Association (Other); Queen's University (Other)
Responsible Party: Sponsor-Investigator, Dr. Denis O'Donnell, Principal Investigator, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: DMED-1926-16
Record Dates: First submitted 2018-01-12; First posted 2018-01-19 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Fentanyl; Albuterol, Ipratropium Drug Combination; Bronchodilator Agents

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fentanyl Citrate (Active Comparator): Single dose, nebulized 100 mcg fentanyl citrate. This is a randomized, double-blind, two-treatment crossover study comparing the effects of a single dose of nebulized 100 mcg fentanyl citrate with a constant fraction of 30% inhaled oxygen to that of a nebulized bronchodilator (Combivent). Treatments will be in randomized order: patients in one study arm will receive fentanyl at the first treatment visit and combivent at the second treatment visit, patients in the other arm will receive Combivent first and fentanyl second.
  Interventions: Drug: Fentanyl Citrate
- Combivent Bronchodilator (Active Comparator): Single dose, nebulized Combivent bronchodilator (0.5 mg ipratropium bromide + 2.5 mg salbutamol). This is a randomized, double-blind, two-treatment crossover study comparing the effects of a single dose of nebulized 100 mcg fentanyl citrate with a constant fraction of 30% inhaled oxygen to that of a nebulized bronchodilator (Combivent). Treatments will be in randomized order: patients in one study arm will receive fentanyl at the first treatment visit and combivent at the second treatment visit, patients in the other arm will receive Combivent first and fentanyl second.
  Interventions: Drug: Combivent

INTERVENTIONS:
Drug: Fentanyl Citrate — 100 mcg fentanyl citrate will be inhaled via nebulizer
  Other Names: Inhaled fentanyl
  Arms: Fentanyl Citrate
Drug: Combivent — 0.5 mg ipratropium bromide + 2.5 mg salbutamol will be inhaled via nebulizer
  Other Names: Bronchodilator
  Arms: Combivent Bronchodilator

SUMMARY:
Activity-related breathlessness (dyspnea) is the dominant symptom and persists despite optimal medical care in as many as 50% of patients with advanced chronic obstructive pulmonary disease (COPD). The objective of this project is to determine the underlying mechanisms of the activity-related breathlessness in patients with advanced COPD. To study the different pathways involved in causing breathlessness, we will compare the effects of two treatments, opiates with oxygen versus bronchodilators, which relieve breathlessness in different ways.

DETAILED DESCRIPTION:
Dyspnea arises during exercise in COPD patients when there is a mismatch between the ventilatory demand (largely dictated by chemical stimuli) and the capacity to respond to that demand (dictated by mechanical/muscular factors). Our preliminary studies have indicated that treatment with opioids in COPD patients can improve activity related dyspnea by reducing central respiratory neural drive and breathing frequency without a significant change in the respiratory mechanics. By contrast, a reduction in exertional dyspnea following inhaled bronchodilators in COPD was mainly related to an improved respiratory mechanics with increased inspiratory capacity, tidal volume, and inspiratory reserve volume etcetera. By comparing the physiological mechanisms of dyspnea relief during the opiate and bronchodilator therapy, we hope to gain new insights into the mechanisms of dyspnea in COPD by selectively manipulating inspiratory neural drive (nebulized opiates) and abnormal respiratory mechanics (nebulized bronchodilators) within the same individuals. As such, the primary objective of this study is to compare the effects of inhaled opiate with oxygen versus bronchodilator treatments on the intensity of dyspnea, electromyographic estimates of inspiratory neural drive and respiratory mechanics and their interactions during a standardized exercise test using a randomized, controlled, crossover design in patients with COPD.

ELIGIBILITY:
Inclusion Criteria:

1. Post-bronchodilator forced expiratory volume in 1 sec (FEV1) 30-79% predicted and FEV1/forced vital capacity (FVC) <70%
2. Clinically stable as defined by no changes in medication dosage or frequency of administration with no exacerbations or hospital admissions in the preceding 6 weeks
3. Male or female ≥40 yrs of age
4. Cigarette smoking history ≥20 pack-years
5. Moderate-to-severe chronic activity-related dyspnea as defined by a modified MRC dyspnea scale ≥2, COPD Assessment Test score ≥10 or Baseline Dyspnea Index focal score ≤6 (47-49)
6. Ability to perform all study procedures and provide/sign informed consent.

Exclusion Criteria:

1. Women of childbearing age who are pregnant or trying to become pregnant
2. Diffusing capacity of the lung for carbon monoxide (DLCO) value of <40 %predicted
3. Active cardiopulmonary disease other than COPD that could contribute to dyspnea and exercise limitation
4. History/clinical evidence of asthma, atopy and/or nasal polyps
5. History of hypercapnic respiratory failure or a clinical diagnosis of sleep disordered breathing
6. History of allergy or adverse response to fentanyl
7. Important contraindications to clinical exercise testing, including inability to exercise because of neuromuscular or musculoskeletal disease(s)
8. Use of daytime oxygen or exercise-induced O2 desaturation to < 80% on room air
9. Body mass index (BMI) <18.5 or ≥35.0 kg/m2
10. Use of antidepressant drugs (i.e., monoamine oxidase inhibitors, serotonin reuptake inhibitors) in previous 2 weeks
11. Use of opioid drugs (e.g., morphine, fentanyl, oxycodone, codeine, etc.) in the previous 4 weeks.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2022-03-21 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Dyspnea intensity measured by the 10-point Borg Scale at a standardized time during cycle exercise test | 10-minutes post-treatment
  The 10-point Borg scale ranges from 0 "nothing at all" to 10 "maximal/extremely strong" and will be used to rate the intensity of dyspnea during exercise: a decrease in this rating signifies an improvement. Dyspnea intensity will be assessed at a standardized time (4-minutes) in both post-treatment constant-load cycle exercise tests.

SECONDARY OUTCOMES:
Diaphragm electromyography (EMGdi) at a standardized time during cycle exercise test | 10-minutes post-treatment
  EMGdi will be used as an index of inspiratory neural drive. Assessments will be compared at a standardized time (4-minutes) during both post-treatment constant-load cycle exercise tests.
Ventilation at a standardized time during cycle exercise test | 10-minutes post-treatment
  Exercise measurements of minute ventilation will be compared at a standardized time (4-minutes) during both post-treatment constant-load exercise tests.
Breathing frequency at a standardized time during cycle exercise test | 10-minutes post-treatment
  Exercise measurements of breathing frequency (respiratory rate) will be compared at a standardized time (4-minutes) during both post-treatment constant-load exercise tests.
Tidal volume at a standardized time during cycle exercise test | 10-minutes post-treatment
  Exercise measurements of tidal volume will be compared at a standardized time (4-minutes) during both post-treatment constant-load cycle exercise tests.
Inspiratory capacity at a standardized time during cycle exercise test | 10-minutes post-treatment
  Exercise measurements of inspiratory capacity will be compared at a standardized time (4-minutes) during both post-treatment constant-load cycle exercise tests.

CONTACTS AND LOCATIONS:
Overall Officials: Denis E O'Donnell, MD, FRCPC, Principal Investigator — Queen's University
Locations (1):
- Respiratory Investigation Unit, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-23): https://cdn.clinicaltrials.gov/large-docs/90/NCT03405090/Prot_SAP_000.pdf